CLINICAL TRIAL: NCT06102629
Title: Understanding the Epigenetic Mechanisms in the Pathophysiology of Polycystic Ovary Syndrome for Efficient Diagnosis and Targeted Therapy
Brief Title: Ovary Syndrome for Efficient Diagnosis and Targeted Therapy
Acronym: PCOS-01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCOS-01
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Laparoscopy; Laparotomy

STUDY DESIGN:
Intervention Model Description: This is a Case control study with two parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100 women undergoing surgery (laparoscopy / laparotomy) with presumed diagnosis of PCOS ( (Experimental): 1. We will take both blood and ovarian tissue samples used to diagnosis.
  2. We will take approximately 3 ml of blood which will be used from the blood sample collected for routine preoperative tests (surgical profile) before their planned surgery or for disease evaluation.
  3. Small tissue samples (from ovary) will be taken from the tissue which is surgically excised as a part of treatment.
  Interventions: Procedure: laparoscopy / laparotomy; Other: NO INTERVENTION
- 100 women undergoing surgery for gynaecological disorder (No Intervention): 1. We will take both blood and ovarian tissue samples used to diagnosis.
  2. We will take approximately 3 ml of blood which will be used from the blood sample collected for routine preoperative tests (surgical profile) before their planned surgery or for disease evaluation.
  3. Small tissue samples (from ovary) will be taken from the tissue which is surgically excised as a part of treatment.

INTERVENTIONS:
Procedure: laparoscopy / laparotomy — 1. We will take both blood and ovarian tissue samples used to diagnosis.
  2. We will take approximately 3 ml of blood which will be used from the blood sample collected for routine preoperative tests (surgical profile) before their planned surgery or for disease evaluation.
  3. Small tissue samples (from ovary) will be taken from the tissue which is surgically excised as a part of treatment.
  Arms: 100 women undergoing surgery (laparoscopy / laparotomy) with presumed diagnosis of PCOS (
Other: NO INTERVENTION — .We will take both blood and ovarian tissue samples used to diagnosis. 2.We will take approximately 3 ml of blood which will be used from the blood sample collected for routine preoperative tests (surgical profile) before their planned surgery or for disease evaluation.
  3. Small tissue samples (from ovary) will be taken from the tissue which is surgically excised as a part of treatment.
  Arms: 100 women undergoing surgery (laparoscopy / laparotomy) with presumed diagnosis of PCOS (

SUMMARY:
OBJECTIVES:

1. Analysis of DNA methyl transferases (DNMT1, DNMT3A and DNMT3B) and Histone deacetylases (HDAC 1,2,3 and SIRTs) polymorphisms (Somatic and germ line variations).
2. Analysis of differential mRNA and protein expression of epigenetic markers in ovarian tissues obtained from PCOS patients.
3. miRNA regulated epigenetic mechanisms in PCOS
4. Epigenetic regulation of endocrine genes in PCOS

DESIGN : A Case Control study.Sample size:200

DETAILED DESCRIPTION:
1. We will take both blood and ovarian tissue samples used to diagnosis.
2. We will take approximately 3 ml of blood which will be used from the blood sample collected for routine preoperative tests (surgical profile) before their planned surgery or for disease evaluation.
3. Small tissue samples (from ovary) will be taken from the tissue which is surgically excised as a part of treatment.

ELIGIBILITY:
Inclusion Criteria:

* All the subjects would be of Indian origin (controls ~100, cases ~100). They would be in their reproductive age (18-45 yrs). Rotterdam consensus would be used to diagnose PCOS and cases will be selected based on it.

Criteria for the diagnosis of PCOS would include oligo-ovulation cycles longer than 35 days or less than 26 days, elevated free testosterone levels (0.5 ng/dl; the cutof level for free testosterone level was the mean±2 SD according to normal levels in controls), oligomenorrhea or amenorrhea.

A Ferriman-Gallwey (FG) score of≥7 would be taken as indicator for the presence of hirsutism. In accordance with the above criteria, polycystic ovary morphology would be determined by transvaginal ultrasonography, which defines PCOS as the presence of 12 or more small (2-9 mm) follicles in each ovary.

Control subjects would have no signs of menstrual dysfunction and their androgen levels should be within the normal range, with normal glucose tolerance, and no family history of hirsutism, type 2 diabetes mellitus, and infertility.

Exclusion Criteria:

* Women with other causes of hyperandrogenism such as hyperprolactinemia, androgen-secreting tumors, Cushing syndrome and nonclassic congenital hyperplasia would be excluded from this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-05 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Analysis of DNA methyl transferases | 3 YEARS
  DNA will be extracted as per the protocol followed routinely in our lab from blood and ovarian tissues.
Evaluate the Analysis of differential mRNA and protein expression of epigenetic markers in ovarian tissues | 3 YEARS
  Total RNA from ovarian tissue will be extracted using TRIzol reagent according to the manufacturer's instructions (Invitrogen Life Technologies) and reverse transcribed in the presence of random hexamers. Quantitative real-time PCR reactions will be carried out in an ABI 7000 Thermal Cycler (Applied Biosystems) to analyse the expression of epigenetic markers including the androgen regulated miRNAs and their downstream targets.

SECONDARY OUTCOMES:
understand miRNA regulated epigenetic mechanisms | 3 YEARS
  The present study would investigate the expression pattern of DNMTs, HDACs, miRNAs and their downstream targets in Ovarian tissues (samples of normal adult ovaries and polycystic ovaries) by western blot and immunohistochemical analysis (IHC).

CONTACTS AND LOCATIONS:
Overall Officials: Shraddha Ramchandani, Principal Investigator — AIG HOSPITALS
Locations (1):
- Dr. Shraddha Ramchandani, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No